CLINICAL TRIAL: NCT03224806
Title: Effect of Fiber Composite-enriched Breads on Glycemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: University of Guelph (Other); Guelph Research and Development Centre, Agriculture and Agri-Food Canada (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GIL-1426
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Glycemic Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wholegrain bread (Other)
  Interventions: Other: Wholegrain bread
- White bread (Other)
  Interventions: Other: White bread
- 15% fiber-rich bread (Other)
  Interventions: Other: 15% fiber-rich bread
- 30% fiber-rich bread (Other)
  Interventions: Other: 30% fiber-rich bread

INTERVENTIONS:
Other: Wholegrain bread — 156.8g wholegrain bread
  Arms: Wholegrain bread
Other: White bread — 122.6g white bread
  Arms: White bread
Other: 15% fiber-rich bread — 139.2g bread made with 15% added wheat bran
  Arms: 15% fiber-rich bread
Other: 30% fiber-rich bread — 166.5g bread made with 30% added wheat bran
  Arms: 30% fiber-rich bread

SUMMARY:
Health organizations recommend fiber-rich and whole-grain foods for healthy diets due to their physiological beneficial effects on human health. But, little information is available between these 2 food categories, i.e. fiber added to foods versus fiber naturally present in foods. The present study investigated the effect of enriching white wheat flour with wheat bran at 2 levels (15 and 30%) to produce 15% fiber-rich bread (15FRB) and 30% fiber-rich bread (30FRB) and compared them with white bread (WB) and whole-grain bread (WGB) in terms of bread quality, palatability, satiety, and glycemic response. Ten healthy subjects were studied on 4 separate days with each subject testing all 4 types of bread. On each test day subjects came to the test center after an overnight fast. After 2 fasting finger-prick blood samples, they ate a portion of one of the breads containing 50g available carbohydrate and had further blood samples at intervals over 2 hours. They also rated their feelings of satiety fasting and at intervals over 2 hours.

DETAILED DESCRIPTION:
Health organizations recommend fiber-rich and whole-grain foods for healthy diets due to their physiological beneficial effects on human health. But, little information is available between these 2 food categories, i.e. fiber added to foods versus fiber naturally present in foods. The present study investigated the effect of enriching white wheat flour with wheat bran at 2 levels (15 and 30%) to produce 15% fiber-rich bread (15FRB) and 30% fiber-rich bread (30FRB) and compared them with white bread (WB) and whole-grain bread (WGB) in terms of bread quality, palatability, satiety, and glycemic response. Ten healthy subjects were studied on 4 separate days with each subject testing all 4 types of bread. On each test day subjects came to the test center after an overnight fast. After 2 fasting finger-prick blood samples 5 minutes apart, they ate a portion of one of the breads containing 50g available carbohydrate and had further blood samples at 15, 30, 45, 60,90 and 120 min after starting to eat. After each blood sample also rated their feelings of satiety on a 7-point scale from extremely hungry to extremely full.

ELIGIBILITY:
Inclusion Criteria:

* Good health

Exclusion Criteria:

* Known history of AIDS, hepatitis, diabetes or a heart condition
* Use of drugs which would increase risk to the subject or affect the results in the opinion of the medical director
* Any condition which would increase risk to the subject or affect the results in the opinion of the medical director
* Individuals who cannot or will not comply with experimental procedures or do not follow safety guidelines.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2014-06-13 (Actual)

PRIMARY OUTCOMES:
Glucose AUC | 2 hours
  Incremental area under the glucose response curve ignoring area below fasting glucose

SECONDARY OUTCOMES:
Satiety AUC | 2 hours
  Incremental area under the satiety response curve
Hydrolysis index | 2 hours
  Incremental area under the hydrolysis curve (amount of glucose released during in-vitro digestion of the breads) expressed as a percentage of that for white bread.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — GI Labs
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No